CLINICAL TRIAL: NCT05324891
Title: Dexmedetomidine Versus Fentanyl for Sedation of Postoperative Mechanically Ventilated Neonates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ms/15.05.90
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fentanyl (Active Comparator): Neonates received fentanyl infusion during postoperative phase.
  Interventions: Drug: Fentanyl
- Dexmedetomidine (Active Comparator): Neonates received dexmedetomidine infusion during postoperative phase.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Infants received dexmedetomidine IV loading dose: 0.5 mcg/kg given over 20 minutes followed by maintenance dose 0.3 µg/kg/hour by infusion over 24 hours.Weaning was done when the patient was about to be extubated or with maximum 5 days after the randomization.
  Arms: Dexmedetomidine
Drug: Fentanyl — Infants received Fentanyl IV continuous infusion: 1µg/ kg /hour. Weaning was done when the patient was about to be extubated or with maximum 5 days after the randomization.
  Arms: Fentanyl

SUMMARY:
Newborn infants experience pain after surgical procedures,prevention and management of pain in neonates is important due to its deleterious consequences. Fentanyl is a widely used analgesic which promotes rapid analgesia,however, is not free of adverse effects including chest wall rigidity, hypothermia, hypotension, respiratory depression and tolerance.Dexmedetomidine is a selective α 2-adrenergic agonist can cause sedation, anxiolysis, analgesia and minimal respiratory depression.Therefore, the objective of the study is to evaluate the safety and efficacy of dexmedetomidine compared to fentanyl in postoperative mechanically ventilated neonates.

DETAILED DESCRIPTION:
A prospective, randomized trial, which was conducted upon neonates who needed postoperative mechanical ventilation in Neonatal Intensive Care Unit, Mansoura University Children's Hospital.The patients were randomized to two groups according to the drug they received for postoperative sedation. The first group received dexmedetomidine infusion and the second group received fentanyl infusion.Our primary outcome was the efficacy of postoperative sedation score, and the secondary outcomes were plasma cortisol level, time to extubation, time to reach 100ml/kg enteral feed, need for adjuvant sedative and skeletal muscle relaxant, length of the hospital stay, side effects of sedative drugs and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Neonates need postoperative ventilation.

Exclusion Criteria:

1. Major congenital cardiovascular anomalies.
2. Chromosomal anomalies.
3. Grade IV intraventricular hemorrhage.
4. Tracheoesophageal fistula with wide gap (distance between proximal and distal end more than two centimeters).

Ages: 1 Hour to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
The efficacy of postoperative sedation according to pain score. | upto five days after surgical intervention
  Assessment of Neonatal Pain, Agitation and Sedation Scale immediately after the operations then every 12 hours till 5 days

SECONDARY OUTCOMES:
Plasma cortisol level | Within 48 hours after surgical intervention
  Plasma as a base line after the operation and another two measures one after 24 hours from the operation and the other after 48 hours
Need of adjuvant analgesics or sedatives | upto five days after surgical intervention
  Infants in both groups received open-label intravenous fentanyl boluses at a dose of 1µg/kg, as adjuvant analgesic when the pain score was more than 3 points. The dose was repeated, based on pain score assessment, at a minimum interval of 2-4 hours. Also, both groups received midazolam bolus at a dose of 0.1 mg/ kg/dose IV as adjuvant sedative in both groups when the patient was agitated.
Need of skeletal muscle relaxant | upto five days after surgical intervention
  Neonates in both groups received Pancuronium at a dose of 0.1 mg/ kg /dose IV as a skeletal muscle relaxant when two boluses of midazolam failed to control agitation
Time to extubation. | upto 21 days postoperative
  Days upon mechanical ventilation
Time to reach 100ml/kg/day enteral feed. | upto 21 days postoperative
  Days to reach 100ml/kg/day enteral feed.
Length of hospital stay. | upto 30 days postoperative
  Days of hospital admission
Mortality | upto 21 days postoperative
  Death
Adverse effects of the sedative drugs | upto seven days after surgical intervention
  Hypotension, bradycardia, chest wall rigidity, feeding intolerance withdrawal signs,re-intubation within 48 hours
Culture-proven sepsis | upto 30 days after surgical intervention

IPD SHARING:
Plan to Share IPD: No